CLINICAL TRIAL: NCT05288270
Title: ROBOCOP (ROBOtic Care of Post-stroke Pain): Study Protocol for a Randomized, Double-blind Trial to Assess Robot-assisted Functional and Motor Recovery and Impact on Post-stroke Pain Development
Brief Title: ROBOtic Care of Post-stroke Pain.
Acronym: Robocop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: S.Anna Rehabilitation Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISA-ROBOCOP
Record Dates: First submitted 2021-11-10; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Robotic rehabilitation; Pain; stroke recovery
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, single center trial will recruit subacute hemiplegic patients of any age with hemiparesis of the arm after stroke. The trial is designed as prospective, exploratory, interventional study without drug. The study does not request the use of drugs. This study protocol follows the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) Checklist.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aramis Group (Experimental): Consecutive patients, admitted to Sant' Anna Institute with diagnosis of stroke after hospital discharge that need motor and cognitive treatment and rehabilitation of neurological diseases.
  Interventions: Device: Aramis
- Conventional Group therapy (Active Comparator): Consecutive patients, admitted to Sant' Anna Institute with diagnosis of stroke after hospital discharge that need motor and cognitive treatment and rehabilitation of neurological diseases.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: Aramis — ARAMIS is composed of two computer-controlled, symmetric and interacting exoskeletons able to compensate the inadequate strength and accuracy of the paretic arm movements, of which it measures residual motor function, and the effect of gravity during rehabilitation. It acts through motion capture of the movements of the unaffected arm. In so doing, the patient is able to replicate the movements of the healthy arm with the paretic arm in synchronous, asynchronous or active-assisted manner. The robot-assisted neurorehabilitation using ARAMIS consists in 60-min sessions for 8 weeks,structured as follows:
  * 1 to 4 weeks: asynchronous exercises of repletion by the paretic arm of basic exercises 20 times for a total of 200 repetitions per session;
  * 5 to 8 weeks: replaced by synchronous exercises (100/session) with active-assisted modality.
  Arms: Aramis Group
Other: Conventional therapy — The control group will receive conventional rehabilitation consisting in passive mobilization of upper and lower limbs, coordination respiratory exercises, cardiovascular conditioning in the setting posture, conditioning in the upright posture, exercises for the trunk control.
  Arms: Conventional Group therapy

SUMMARY:
In agreement to the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) recommendations that support the importance of physical functioning as core outcome for pain this randomized, double-blind, controlled clinical trial will be the pilot forming the rational basis for the assessment of the efficacy in the use of Robotic rehabilitation system to prevent chronic post stroke pain development. In fact, according to working hypothesis, proprioceptive inputs with high-intensive bilateral movement training of the hemiplegic arm can improve recovery and plasticity, thus preventing chronic post-stroke pain from occurring within the 3-6 months following stroke.

DETAILED DESCRIPTION:
Stroke is one of the most frequent causes of death and disability worldwide. It is accompanied by impaired motor function of the upper extremities in over 69% of patients up to hemiplegia in the following 5 years in 56% of cases. This condition often is characterized by chronic post-stroke pain, difficult to manage and further worsening the patients' quality of life. Post-stroke pain occurs within 3-6 months and aberrant neuroplasticity in the first 3-4 weeks is implicated in its development. Robot-assisted neurorehabilitation using the Automatic Recovery Arm Motility Integrated System (ARAMIS) has proven efficacy in motor function recovery exploiting the movements and the strength of the unaffected arm to drive correct brain re-arrangement. Therefore, the rationale of the ROBOCOP (ROBOtic Care of Post-stroke pain) randomized, double-blind trial for the assessment of the impact of robot-assisted functional and motor recovery on post-stroke pain development is based on the prevention of anomalous plasticity and, hopefully, on the recovery of connectivity in the injured area.

To this aim, a total of 118 patients with hemiplegic arm due to stroke will be enrolled and randomly allocated with 1:1 ratio to ARAMIS or conventional neurorehabilitation group. After a baseline screening at hospital discharge during subacute period, ARAMIS or conventional rehabilitation will be performed for 8 weeks. The primary endpoint will consist in improvement of the Upper Extremity Subscale of the Fugl-Meyer Motor Assessment (FMA-UE), for the body functions of the upper extremity section domain; the Action Research Arm Test (ARAT) scores at 1, 2, 3 and 6 months after stroke. The secondary endpoints include no worsening of pain Visual Analogue Scale (VAS) and improvement of Barthel Index (BI) for activities of daily living and of Frenchay activities index (FAI) for physical activity, as well as improvement of magnetic resonance imaging (MRI) and electroencephalographic (EEG) parameters This is the first clinical trial investigating the efficacy of robot-assisted neurorehabilitation using ARAMIS on brain plasticity and re-organization and on post-stroke pain prevention. This study could remarkably improve the quality of life of stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Stroke-related hemiplegic arm;
* Hemiplegic subacute patients of any age at hospital discharge after stroke with functional magnetic resonance imaging (fMRI) scan of the area affected.

Exclusion Criteria:

Bilateral impairment;

* Presence of aphasia;
* Presence of cognitive impairment;
* Stroke diagnosis without occurrence of hemiparesis of the upper limb.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Assessment - upper extremity (FMA-UE) | up to 6 months after the admission assessment.
  Improvement of Fugl-Meyer Motor Assessment (FMA-UE) scores. The score may range from 0 to 115. A higher score indicates better recovery
Action Research Arm Test (ARAT)- Motor recovery scale | up to 6 months after the admission assessment.
  Improvement of Action Research Arm Test (ARAT) scores. Scores on the ARAT may range from 0-57 points, with a maximum score of 57 points indicating better performance
Visual Analogue Scale (VAS) - Pain reduction | up to 6 months after the admission assessment.
  No worsening of Visual Analogue Scale (VAS). Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in patients who described their pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Barthel Index (BI) | up to 6 months after the admission assessment.
  Improvement of Barthel Index (BI). Scores on the BI may range from 0-100 points, with a maximum score of 100 points. Score from 80 to 100 indicates that the patient should be able to live indipendently

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual partecipant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after the end of the study
Access Criteria: Data access request will be reviewed by an internal audit committee in conjunction with a panel of university experts

REFERENCES:
- [Result] Cerasa A, Pignolo L, Gramigna V, Serra S, Olivadese G, Rocca F, Perrotta P, Dolce G, Quattrone A, Tonin P. Exoskeleton-Robot Assisted Therapy in Stroke Patients: A Lesion Mapping Study. Front Neuroinform. 2018 Jul 17;12:44. doi: 10.3389/fninf.2018.00044. eCollection 2018. PMID 30065642
- [Result] Pignolo L, Serra S, Basta G, Carozzo S, Arcuri F, Pignataro LM, Ciancarelli I, Tonin P, Cerasa A. Data on a new neurorehabilitation approach targeting functional recovery in stroke patients. Data Brief. 2019 Oct 28;27:104685. doi: 10.1016/j.dib.2019.104685. eCollection 2019 Dec. PMID 31737755
- [Result] Pignolo L. Robotics in neuro-rehabilitation. J Rehabil Med. 2009 Nov;41(12):955-60. doi: 10.2340/16501977-0434. PMID 19841823
- [Result] Calabro RS, Filoni S, Billeri L, Balletta T, Cannavo A, Militi A, Milardi D, Pignolo L, Naro A. Robotic Rehabilitation in Spinal Cord Injury: A Pilot Study on End-Effectors and Neurophysiological Outcomes. Ann Biomed Eng. 2021 Feb;49(2):732-745. doi: 10.1007/s10439-020-02611-z. Epub 2020 Sep 11. PMID 32918105
- [Result] Calabro RS, Pignolo L, Muller-Eising C, Naro A. Pain Perception in Disorder of Consciousness: A Scoping Review on Current Knowledge, Clinical Applications, and Future Perspective. Brain Sci. 2021 May 20;11(5):665. doi: 10.3390/brainsci11050665. PMID 34065349
- [Result] Colizzi L, Lidonnici A, Pignolo L. The ARAMIS project: a concept robot and technical design. J Rehabil Med. 2009 Nov;41(12):1011-101. doi: 10.2340/16501977-0407. PMID 19841834
- [Result] Gandolfi M, Vale N, Posteraro F, Morone G, Dell'orco A, Botticelli A, Dimitrova E, Gervasoni E, Goffredo M, Zenzeri J, Antonini A, Daniele C, Benanti P, Boldrini P, Bonaiuti D, Castelli E, Draicchio F, Falabella V, Galeri S, Gimigliano F, Grigioni M, Mazzon S, Molteni F, Petrarca M, Picelli A, Senatore M, Turchetti G, Giansanti D, Mazzoleni S; Italian Consensus Conference on Robotics in Neurorehabilitation (CICERONE). State of the art and challenges for the classification of studies on electromechanical and robotic devices in neurorehabilitation: a scoping review. Eur J Phys Rehabil Med. 2021 Oct;57(5):831-840. doi: 10.23736/S1973-9087.21.06922-7. Epub 2021 May 27. PMID 34042413
- [Result] Paolucci S, Iosa M, Toni D, Barbanti P, Bovi P, Cavallini A, Candeloro E, Mancini A, Mancuso M, Monaco S, Pieroni A, Recchia S, Sessa M, Strambo D, Tinazzi M, Cruccu G, Truini A; Neuropathic pain special interest group of the Italian Neurological Society. Prevalence and Time Course of Post-Stroke Pain: A Multicenter Prospective Hospital-Based Study. Pain Med. 2016 May;17(5):924-30. doi: 10.1093/pm/pnv019. Epub 2015 Dec 14. PMID 26814255
- [Result] Scuteri D, Mantovani E, Tamburin S, Sandrini G, Corasaniti MT, Bagetta G, Tonin P. Opioids in Post-stroke Pain: A Systematic Review and Meta-Analysis. Front Pharmacol. 2020 Nov 27;11:587050. doi: 10.3389/fphar.2020.587050. eCollection 2020. PMID 33424596
- [Result] Scuteri D, Corasaniti MT, Tonin P, Bagetta G. Eptinezumab for the treatment of migraine. Drugs Today (Barc). 2019 Nov;55(11):695-703. doi: 10.1358/dot.2019.55.11.3069864. PMID 31840684
- [Result] Scuteri D, Rombola L, Morrone LA, Bagetta G, Sakurada S, Sakurada T, Tonin P, Corasaniti MT. Neuropharmacology of the Neuropsychiatric Symptoms of Dementia and Role of Pain: Essential Oil of Bergamot as a Novel Therapeutic Approach. Int J Mol Sci. 2019 Jul 6;20(13):3327. doi: 10.3390/ijms20133327. PMID 31284573
- [Result] Dolce G, Lucca LF, Pignolo L. Robot-assisted rehabilitation of the paretic upper limb: rationale of the ARAMIS project. J Rehabil Med. 2009 Nov;41(12):1007-101. doi: 10.2340/16501977-0406. PMID 19841833
- [Result] Pignolo L, Lucca LF, Basta G, Serra S, Pugliese ME, Sannita WG, Dolce G. A new treatment in the rehabilitation of the paretic upper limb after stroke: the ARAMIS prototype and treatment protocol. Ann Ist Super Sanita. 2016 Apr-Jun;52(2):301-8. doi: 10.4415/ANN_16_02_25. PMID 27364408
- [Result] Cramer SC. Functional imaging in stroke recovery. Stroke. 2004 Nov;35(11 Suppl 1):2695-8. doi: 10.1161/01.STR.0000143326.36847.b0. Epub 2004 Sep 23. PMID 15388899
- [Result] Lee J, Park E, Lee A, Chang WH, Kim DS, Kim YH. Recovery-related indicators of motor network plasticity according to impairment severity after stroke. Eur J Neurol. 2017 Oct;24(10):1290-1299. doi: 10.1111/ene.13377. Epub 2017 Aug 18. PMID 28833921
- [Result] Ustinova KI, Goussev VM, Balasubramaniam R, Leven MF. Disruption of coordination between arm, trunk, and center of pressure displacement in patients with hemiparesis. Motor Control. 2004 Apr;8(2):139-59. doi: 10.1123/mcj.8.2.139. PMID 15118199